CLINICAL TRIAL: NCT06309056
Title: Evaluating the Effectiveness of Neuromuscular Electrical Stimulation for Children With Dysphagia: A Pilot Study
Brief Title: Neuromuscular Electrical Stimulation for Children With Dysphagia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Sam Daniel, Pediatric Otolaryngologist, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP-05-2024-3903
Record Dates: First submitted 2024-02-29; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Dysphagia
Keywords: neuromuscular electrical stimulation; pediatric dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Patients being followed at the Lethbridge-Layton-Mackay Rehabilitation Centre Salivation Management Clinic and the Dysphagia and Feeding Disturbance Clinic who meet inclusion criteria will be recruited. If caregivers/participants consent to the study, they will be enrolled in the intervention arm. Any potentially eligible participant who declines to participate in the study will be recruited as a control group. These participants will complete the questionnaires at the same timepoints as the interventional group and data from the medical charts will be included in the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Interventional Group (Experimental)
  Interventions: Device: VitalStim
- Control Group (No Intervention)

INTERVENTIONS:
Device: VitalStim — VitalStim is a device that provides neuromuscular electrical stimulation. It will be applied on muscles related to swallowing to stimulate muscle contraction.
  Arms: Interventional Group

SUMMARY:
This study aims to measure if using neuromuscular electrical stimulation (NMES) effectively improves swallowing, drooling (if applicable), feeding ability, physical growth and quality of life in children with severe dysphagia. This pilot study is for children aged over 18 months old with dysphagia. It aims to investigate a new approach to help children improve their swallowing function. Some published studies have shown that electrical stimulation to muscles involved in swallowing may help children with dysphagia.

In this pilot study, NMES will be used. This procedure delivers electrical stimulation to make participants' muscles contract. Electrodes are placed on the skin, over the muscles that help with swallowing, and an electric current is delivered through wires which are connected to a small machine. The current is controlled through a small, handheld device. NMES will be applied to muscles involved in eating, drinking and swallowing. NMES will be applied to the participant alongside their regular treatment. No medications or treatments will be added, modified or discontinued as part of this study.

The overall duration of the study per participant will last a total of nine months. For the first three months, the participant will receive the NMES twice a week. There will be no interventions or follow-up appointments scheduled for the following 6 months. Then, there will be a final follow-up meeting 9 months following the start of the intervention to evaluate for lasting changes.

DETAILED DESCRIPTION:
The proposed study will consist of a sample size of 10 to 20 children over 18 months diagnosed with oropharyngeal dysphagia, as confirmed by fiberoptic endoscopic evaluation of swallowing (FEES) or videofluoroscopic swallowing study (VFSS). Participants will be recruited at the Lethbridge-Layton-Mackay Rehabilitation Centre Salivation Management Clinic and the Dysphagia and Feeding Disturbance Clinic.

The sample size is based on the number of children who are followed at this clinic who would likely meet the inclusion criteria for this study. It is also based on the availability of human resources.

Participants will be recruited at the Lethbridge-Layton-Mackay Rehabilitation Centre Salivation Management Clinic and the Dysphagia and Feeding Disturbance Clinic. Any instrumental swallowing examination performed up to one year before initiating interventions, at any point during the study, and up to one year following the completion of the interventions, will be retrieved.

VitalStim pediatric electrodes will be placed depending on the impairment causing the child's dysphagia. Electrodes will only be placed on intact skin. No current channels will be placed on a surgical incision or through indwelling foreign material such as tracheostomy, staples or sutures. Current will be applied at the highest tolerated intensity, between 2-25 milliamps. As per the individualized nature of this intervention, the intensity will be individualized per patient and per session. A therapeutic intensity range will be determined by assessing for two or more of the following signs: a change in the audible quality of swallow, description of grabbing/pulling, triggered swallowing, better swallowing than without NMES as evaluated by the clinician (stronger muscles involved in swallowing by palpation, decrease in drooling, improved lip closure, decreased signs of aspiration, ability to swallow a higher quantity of food, ability to swallow food of better consistency), sitting up straight, reaching for electrodes or change of voice. The other parameters will be based on the VitalStim protocol: frequency 80 pps, phase duration 300 microseconds and duty cycle 57:1.

Each session will last up to 45 minutes, as tolerated by the child, twice weekly, for three months. The overall duration of the study will last nine months. For the first three months, the participant will receive the intervention twice a week. There will then be a final follow-up meeting six months after the final intervention. There will be a total of 25 sessions. At the first session, participants and their parent/caregiver will complete four questionnaires evaluating the child's feeding ability, the child's drooling, the child's overall quality of life and the impact and stress that feeding difficulties have on the child's parent. Each questionnaire will take approximately 5 minutes to complete. If the child has a developmental age of 4 or below, the parent/caregiver will complete all the questionnaires. If the child has a developmental age of 5 or older, they will complete one questionnaire by themselves, and the others will be completed by the parent/caregiver. Also, the child will be measured and weighed. These parameters will be repeated at the final intervention session (week 12) and six months later (week 36).

ELIGIBILITY:
Inclusion Criteria:

* Children with oropharyngeal dysphagia
* Children aged over 18 months
* Children with the ability to swallow
* Children and their caregiver(s) have a good cooperation and motivation
* Families are able and willing to participate in the study
* Children and their families understand and communicate in English or French

Exclusion Criteria:

* Children with esophageal dysphagia
* Children without dysphagia
* Children who are unable to swallow or who are unaware of having liquid/food in their mouths
* Children with solely anatomical etiologies of dysphagia such as obstructing tumors
* Children aged less than 18 months, and adults 18 years of age and older
* Children and their families do not communicate in English or French
* Children with neuromuscular diagnoses
* Children with vagal nerve stimulators
* Children with cancerous lesions, inflamed or infected skin or skin eruptions in the treatment area

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Feeding Intake - Functional Oral Intake Scale | 12 weeks, 36 weeks
  Feeding intake will be assessed using the Functional Oral Intake Scale. This scale assesses one's ability to tolerate oral intake of various consistencies. This scale is scored from 0 to 7. A higher score indicates a better outcome.

SECONDARY OUTCOMES:
Penetration and Aspiration Scale | 12 weeks, 36 weeks
  Penetration and aspiration will be assessed using functional endoscopic swallowing studies or videofluoroscopic swallowing studies, if available as part of the participant's regular treatment. This scale is scored from 0 to 8. A lower score indicates a better outcome.
Quality of Life - Pediatric Quality of Life Inventory 4.0 Generic Core Scale for Toddlers, Young Children, Children 8-12 years old OR Teenagers. | 12 weeks, 36 weeks
  The quality of life of children will be assessed using the Pediatric Quality of Life Inventory using the form specific to the age of the participant. The score is from 0 to 84 (toddlers), 0 to 92 (young children), 0 to 92 (children 8-12) and 0 to 60 (teenagers). A lower score indicates a better outcome.
Body Mass Index (kg/m^2) | 12 weeks, 36 weeks
  Height in m^2 and weight in kilograms will be obtained to measure the body mass index. A higher score indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sam Daniel, MD, Principal Investigator — McGill University

IPD SHARING:
Plan to Share IPD: No
It is undecided.